CLINICAL TRIAL: NCT03989609
Title: ROle of Dexmedetomidine in Modifying Immune Paralysis In Patient With Septic Shock: Randomized Controlled Trial (RODIS Trial)
Brief Title: Dexmedetomidine in Modifying Immune Paralysis In Patient With Septic Shock
Acronym: RODIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Elayashy Mohamed Ahmed Hassan, Lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-5-2019
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): patients will receive dexmedetomidine as sedative
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Midazolam (Active Comparator): patients will receive midazolam as sedative
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — Dexmedetomidine infusion will be started at 0.1 µg.kg-1.hr-1 and will be adjusted by 0.1 µg.kg-1.h-1 to a maximum of 0.5 µg/kg/h,
  Arms: Dexmedetomidine Group
Drug: Midazolam — midazolam will be started at 1 mg.h-1 (3 mL.hr-1) and adjusted by 1 mg.h-1 to a maximum of 5 mg.h-1 (15 mL.h-1).
  Arms: Midazolam

SUMMARY:
in this study the investigators aim to assess the role of using dexmedetomidine as sedative in septic shock patients in comparison with midazolam. The investigators aim to assess the effect on immune response and inflammatory mediators and effect on vasopressors.

DETAILED DESCRIPTION:
Sedation protocol All patients will receive analgesia with fentanyl at ﬁxed dose of 0.5 µg.kg.hr-1. Each patient will receive the study drug within 6 hours after ICU admission. Depth of sedation will be assessed using Richmond Agitation and Sedation Scale (RASS) scores (6), which range from -5 (unarousable) to +4 (combative). Study treatments will be infused without loading dose. Group I patients will have dexmedetomidine (4 µg.mL-1) and group II patients will have midazolam (0.33 mg.mL-1). Both drugs will be prepared in 0.9% sodium chloride in 50-mL syringe. Both the agents will be titrated to maintain the RASS in a range of -3 to -1. Dexmedetomidine infusion will be started at 0.1 µg.kg-1.hr-1 and will be adjusted by 0.1 µg.kg-1.h-1 to a maximum of 0.5 µg/kg/h, while midazolam will be started at 1 mg.h-1 (3 mL.hr-1) and adjusted by 1 mg.h-1 to a maximum of 5 mg.h-1 (15 mL.h-1). All infusions will be adjusted by increments of 3 mL/hr-1. Patients in either group not adequately sedated by study drug titration will receive a bolus dose of fentanyl 0.5-1 µg.kg. Assessment of RASS score will be performed every 2 hours and prior to any dose of rescue therapy. The study drugs will be infused for 24 hours and after that the choice of sedation will be determined according to preference of attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* All mechanically ventilated patients who will be clinically suspected of having septic shock defined by infusion of at least one vasopressor and lactate > 2.0 mmol/l (5)

Exclusion Criteria:

* Age < 18 years old
* Pregnant patient
* Source of sepsis not controlled
* Acute hepatitis or severe liver disease (Child-Pugh class C)
* Left ventricular ejection fraction less than 30%
* Heart rate less than 50 beats/min
* Second or third degree heart block
* Systolic pressure < 90 mmHg despite of infusion of 2 vasopressors.
* Psychological illness or severe cognitive dysfunction
* Patients who are allergic to dexmedetomidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Change in CD42/CD14 | 24 hours after start of study drugs infusion
  Expression of CD42/CD14 will be measured by flow cytometry

SECONDARY OUTCOMES:
effect on HLA-DR/CD14 | Baseline before start of drug then 6, 12 and 24 hour after drug
  Expression of HLA-DR/CD14 will be measured by flow cytometry
TNFα | Baseline before start of drug then 6, 12 and 24 hour after drug
  Expression of tumor necrosis factor (TNFα) will be measured by flow cytometry
IL10 | Baseline before start of drug then 6, 12 and 24 hour after drug
  Interleukin 10 will be measured by flow cytometry
KIM-1 level | Baseline before start of drug and 24 hour after drug
  kidney injury molecule 1
number of participants that will die within 28 days | within 28 dyas
  mortality within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Mukhtar, M,D, Study Director — kasralainy faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy Hospital , Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biswas SK, Lopez-Collazo E. Endotoxin tolerance: new mechanisms, molecules and clinical significance. Trends Immunol. 2009 Oct;30(10):475-87. doi: 10.1016/j.it.2009.07.009. Epub 2009 Sep 24. PMID 19781994
- [Background] Yeaman MR. Platelets in defense against bacterial pathogens. Cell Mol Life Sci. 2010 Feb;67(4):525-44. doi: 10.1007/s00018-009-0210-4. Epub 2009 Dec 15. PMID 20013024
- [Background] Miranda ML, Balarini MM, Bouskela E. Dexmedetomidine attenuates the microcirculatory derangements evoked by experimental sepsis. Anesthesiology. 2015 Mar;122(3):619-30. doi: 10.1097/ALN.0000000000000491. PMID 25313879
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Derived] Elayashy M, Elsayed EA, Mukhtar AM, Kasem S, Elmetwally SA, Habib S, Abdelfattah W, Ghaith D, Hussein A. Role of dexmedetomidine in modifying immune paralysis in patients with septic shock: randomized controlled trial. Intensive Care Med Exp. 2023 Sep 4;11(1):59. doi: 10.1186/s40635-023-00542-2. PMID 37665397